CLINICAL TRIAL: NCT03964441
Title: ANDDI-PRENATOME - Feasibility Study for a " Fast " Pangenomic High Throughput Sequencing Analysis in Prenatal Diagnosis
Acronym: AnddiPrenatome
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: THAUVIN AnDDI rares 2018
Record Dates: First submitted 2019-05-22; First posted 2019-05-28 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Prenatal; Genome-wide High Throughput Sequencing
MeSH Terms: interventions — Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- control: fetus with at least 2 ultrasound abnormalities and both parents
  Interventions: Biological: Invasive fetal sampling, blood sampling of mother and father; Other: Parent interviews (optional organizational study); Other: parent questionnaire (optional organizational study)
- comparison: fetus with at least 2 ultrasound abnormalities with ES diagnosis on invasive fetal sampling
  Interventions: Biological: Invasive fetal sampling, blood sampling of mother and father; Biological: blood sampling from the mother to recover the circulating cell free fetal DNA; Other: Parent interviews (optional organizational study); Other: parent questionnaire (optional organizational study)
- professional: obstetrician, midwife, geneticist, biologist
  Interventions: Other: professional interviews (optional organizational study); Other: Focus group for professionals (optional organizational study)

INTERVENTIONS:
Biological: Invasive fetal sampling, blood sampling of mother and father — to perform an exome sequencing analysis in trio
  Groups: comparison; control
Biological: blood sampling from the mother to recover the circulating cell free fetal DNA — to perform a sequencing analysis of the genome of circulating free fetal DNA
  Groups: comparison
Other: Parent interviews (optional organizational study) — Interview with a sociologist or psychologist to explore perceptions of ES and the impact of the results, expectations regarding certain types of results not currently available, the emotional situation, and position regarding the continuation of the pregnancy At 4 different times: at inclusion, at the time of the CGA-array results, at the time of the ES results and at a distance from the ES results
  Groups: comparison; control
Other: parent questionnaire (optional organizational study) — To evaluate the experience, perceptions, the impact of the analyses on the decision, satisfaction and concerns regarding the ES and its results, opinions on certain types of results not currently available, as well as anxiety and possible psychological distress At 4 different points in time: at inclusion, at the delivery of the CGA-array results, at the delivery of the ES results and at a distance from the delivery of the ES results
  Groups: comparison; control
Other: professional interviews (optional organizational study) — interview to understand how the decision is formed
  Groups: professional
Other: Focus group for professionals (optional organizational study) — interview to specify whether variants of unknown significance) VUS will potentially be returned to the clinicians, or even to the patient via the clinician.
  Groups: professional

SUMMARY:
Prenatal diagnosis of genetic diseases is a real medical challenge. The discovery of antenatal abnormalities on ultrasound is frequent (5 to 10% of pregnancies), and when an abnormalities is seen on ultrasound, it raises the possibility of an underlying developmental anomaly. Currently, in France, when abnormalities are discovered with an ultrasound scan, the etiological diagnosis is based on additional imaging tests (cerebral MRI, 3D bone tomography, fetal CT, fetal CT) or diagnostic tests such as invasive chorionic villus sampling, amniocentesis or fetal blood for infectious, metabolic, immunological and genetic investigations (standard karyotype, FISH (fluorescence in situ hybridization) for the rapid detection of aneuploidy, Chromosome Analysis on DNA Chip (ACPA or CGH-array) and possible sequencing of targeted genes when they are available within a time frame compatible with pregnancy). NIPT (Non-invasive prenatal testing) on cell free fetal DNA circulating in maternal blood has more limited indications, allowing, from an early stage of pregnancy, the determination of fetal sex and fetal rhesus factor and the search for aneuploidy.

However, establishing an etiological diagnosis during pregnancy has many benefits for the parents: clarifying the cause, obtaining a more precise prognosis to determine future management and outcome of the pregnancy, and establishing the risks of recurrence.

Over the past decade, medical genetics has undergone a real technological revolution, leading to the development of high throughput genome-wide, exome (ES) and genome (GS) sequencing. However, few countries have currently embarked on ES/GS in prenatal care, due to the constraints of time and the difficulty of interpreting genomic data when the clinical data is limited to antenatal imaging data.

In 2016, France launched the France Medicine Genomics 2025 Plan (PFMG2025) to deploy GS, particularly in the diagnosis of rare diseases. It is thus becoming essential to define the modalities of prescription of this testing, in particular during prenatal diagnosis. In parallel, from the first publications, the applications of genomic analysis on circulating fetal DNA seem to be able to extend to genome sequencing for research of SNVs responsible for developmental diseases.

The AnDDI-rares health network therefore proposes this ANDDI-PRENATOME pilot project to study the feasibility of a "rapid" analysis of ES in prenatal diagnosis from 61 fetuses with ultrasound abnormalities, as a first step before considering future cost-effectiveness (PRME) or care system performance (PREPS) studies in conjunction with the PFMG2025.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with antenatal discovery of at least two obstetric ultrasound abnormalities (2 major malformations, or 1 major malformation and 1 minor malformation, or 1 isolated malformation with a high probability of a genetic condition) : who undergo invasive antenatal sampling for CGH-array diagnosis ; who has already had an invasive antenatal sampling for the diagnosis of CGH-array and for which the fetal CGH-array has been found to be normal (sufficient fetal DNA or amniotic fluid should be available to allow exome sequencing to be performed without further amniotic fluid puncture).
* Pregnant woman and father aged 18 years or more
* Written consent provided by the pregnant woman and the father of the fetus
* Possibility of sufficient fetal specimen (amniotic fluid or fetal blood) to collect an additional sample for the pilot project
* Possibility of sampling the pregnant woman and the father of the foetus (peripheral blood)
* Pregnant woman and father of the fetus able to understand the study

Pilot Organizational Study:

In addition to the inclusion & exclusion criteria of the main study:

* Pregnant woman and biological father of fetus who provided oral consent to be interviewed
* Professionals (obstetrician, midwife, geneticist, biologist) agreeing to be interviewed

Exclusion Criteria:

* Diagnostic hypothesis considered highly probable that can be confirmed by an available molecular or cytogenetic test with a lower cost than ES (e. g. 22q11 microdeletion) or high suspicion of fetal infection (e. g. toxoplamosis seroconversion)
* Refusal of pregnant woman or father of fetus to participate in the study
* Pregnancy earlier than 15 weeks of amenorrhea or later than 34 weeks of amenorrhea
* Pregnant woman and father of the foetus not covered by the national health insurance system
* Pregnant woman and/or father of the fetus under partial judicial protection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women with antenatal discovery of at least two obstetrical ultrasound abnormalities
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Time required to return ES results to patients and their families in a context prenatal diagnosis | Through study completion, an average of 12 months
number of discrepancies between ES and WGS | Through study completion, an average of 12 months

SECONDARY OUTCOMES:
Questionnaire to understand the expectations of couples and their a priori perception of ES | Through study completion, an average of 12 months
  To define feelings and to know better how couples perceive ES and its implications and in particular the risk of discovery of VUS (variants of unknown significance) and ID (incidental data).
Questionnaire to evaluate the organization of health professionals involved in the decision-making process | Through study completion, an average of 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Tran Mau-Them F, Delanne J, Denomme-Pichon AS, Safraou H, Bruel AL, Vitobello A, Garde A, Nambot S, Bourgon N, Racine C, Sorlin A, Moutton S, Marle N, Rousseau T, Sagot P, Simon E, Vincent-Delorme C, Boute O, Colson C, Petit F, Legendre M, Naudion S, Rooryck C, Prouteau C, Colin E, Guichet A, Ziegler A, Bonneau D, Morel G, Fradin M, Lavillaureix A, Quelin C, Pasquier L, Odent S, Vera G, Goldenberg A, Guerrot AM, Brehin AC, Putoux A, Attia J, Abel C, Blanchet P, Wells CF, Deiller C, Nizon M, Mercier S, Vincent M, Isidor B, Amiel J, Dard R, Godin M, Gruchy N, Jeanne M, Schaeffer E, Maillard PY, Payet F, Jacquemont ML, Francannet C, Sigaudy S, Bergot M, Tisserant E, Ascencio ML, Binquet C, Duffourd Y, Philippe C, Faivre L, Thauvin-Robinet C. Prenatal diagnosis by trio exome sequencing in fetuses with ultrasound anomalies: A powerful diagnostic tool. Front Genet. 2023 Mar 23;14:1099995. doi: 10.3389/fgene.2023.1099995. eCollection 2023. PMID 37035737
- [Derived] Thauvin-Robinet C, Garde A, Delanne J, Racine C, Rousseau T, Simon E, Francois M, Moutton S, Sylvie O, Quelin C, Morel G, Goldenberg A, Guerrot AM, Vera G, Gruchy N, Colson C, Boute O, Abel C, Putoux A, Amiel J, Guichet A, Isidor B, Deiller C, Wells C, Rooryck C, Legendre M, Francannet C, Dard R, Sigaudy S, Bruel AL, Safraou H, Denomme-Pichon AS, Nambot S, Asensio MH, Binquet C, Duffourd Y, Vitobello A, Philippe C, Faivre L, Tran-Mau-Them F, Bourgon N. Prenatal exome sequencing, a powerful tool for improving the description of prenatal features associated with genetic disorders. Prenat Diagn. 2024 Sep;44(10):1179-1197. doi: 10.1002/pd.6623. Epub 2024 Aug 13. PMID 39138116